CLINICAL TRIAL: NCT02081612
Title: Comparison of Weight Loss Among Early Stage Breast Cancer Patients Post Chemotherapy: Nutrition Education in Combination With Weight Loss Acupuncture Vs. Nutrition Education Alone
Brief Title: Comparison of Nutrition Education Alone or With Acupuncture for Weight Loss in Breast Cancer Patients Post-Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Tiersten, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 14-0001
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nutrition Assessment; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition Education (Active Comparator): Educational weight management group sessions alone
  Interventions: Behavioral: Nutrition Education
- Nutrition Education Plus Acupuncture (Active Comparator): Educational weight management group sessions in addition to weight loss acupuncture
  Interventions: Behavioral: Nutrition Education; Procedure: Acupuncture

INTERVENTIONS:
Behavioral: Nutrition Education — 12 educational weight management group session each addressing a different weight loss topic
Procedure: Acupuncture — 12 weight loss acupuncture session using both body and auricular points.
  Arms: Nutrition Education Plus Acupuncture

SUMMARY:
This study looks at the benefit of adding acupuncture to nutrition education for weight loss in women with early stage breast cancer post-chemotherapy.

DETAILED DESCRIPTION:
Obesity and weight gain are significant concerns for breast cancer survivors. Given the adverse consequences of weight gain after diagnosis, continued efforts to identify appropriate weight management interventions aimed at promoting overall health and long term survivorship are needed. In this study, the investigators will examine whether adding acupuncture to a nutrition education program for weight loss could improve short and long term weight loss among breast cancer survivors post treatment with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Woman with a diagnosis of breast cancer, stage I, II, or III
* Age ≥ 18
* ECOG performance status ≤ 1
* Received treatment for breast cancer, and treatment must have been completed at least 2 weeks prior to enrollment in trial, but no longer than 1 year post-treatment.
* BMI ≥ 30
* Adequate bone marrow and organ function as determined by the consenting/enrolling investigator
* Signed informed consent
* Any receptor status
* Participant is willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits, and examinations

Exclusion Criteria:

* Current chemotherapy or radiation therapy. Participants in study may still be receiving hormone or Herceptin treatment.
* Diagnosis of metastatic breast cancer
* Participation in other diet-based weight loss programs (ie. Patient should not be currently enrolled in Weight Watchers, Jenny Craig, Nutrisystem, etc.)
* Current use of commercial or natural/herbal weight loss supplements
* Major surgery within 1 month of starting study program and patients must have recovered from any effects of major surgery
* Other malignancies within the past three years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Personal history of an eating disorder
* Other serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection (including uncontrolled HIV, Hepatitis B or C), or any psychiatric disorder that prohibits obtaining informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03-06 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 24 weeks

SECONDARY OUTCOMES:
Maintenance of weight loss | 24 months
Recurrence of breast cancer | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States